CLINICAL TRIAL: NCT05096260
Title: Community-Centered Interventions for Improved Vaccine Uptake for COVID-19 (CIVIC): Getting to Yes, Michigan! (G2YMI)
Brief Title: Getting to Yes, Michigan! (G2YMI)
Acronym: G2YMI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Ken Resnicow, Professor, Health Behavior & Health Education, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: G2YMI; 1R01MD016867-01 (NIH)
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: COVID-19 Vaccines; COVID-19 Pandemic
Keywords: COVID-19 Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Individually randomized control design: control participants will receive the intervention after completion of the follow-up survey (at six months).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Enrolled study participants receive Motivational Interviewing based SMS/MMS messages to increase COVID-19 vaccine uptake, and complete Baseline and Follow-up surveys.
  Interventions: Behavioral: Motivational Interviewing based SMS/MMS and web content
- Control (No Intervention): Enrolled study participants receive a simple website and complete a Baseline and Follow-up survey, after which they will receive the interventional Motivational Interviewing based SMS/MMS messages to increase COVID-19 vaccine uptake.

INTERVENTIONS:
Behavioral: Motivational Interviewing based SMS/MMS and web content — Our primary framework that will guide the web content is Self-Determination Theory (SDT). SDT differentiates between autonomous (conscious choice and are personally relevant) and controlled behavioral regulation (performed due to pressure or coercion by external or internal forces). Messages that enhance autonomy and perceived competence and are consistent with a person's values and goals will be more effective in changing behavior than messages focusing on external rewards. To link vaccination to broader values and goals, participants will select 3-4 goals from approximately 20 values/goals. Individually tailored messages will link each of these values to vaccination. We will also tailor testimonials based on member values and communication style preference.
  Arms: Intervention

SUMMARY:
This study entitled Community-Centered Interventions for Improved Vaccine Uptake for COVID-19 (CIVIC): Getting to Yes, Michigan!, is designed to increase vaccine uptake among populations that experience COVID-19 related disparities. The investigators will focus on the four counties within Michigan where a disproportionate burden of COVID-19 is within African Americans and Latinx communities, i.e., Wayne, Genesee, Kent and Washtenaw Counties. Using a community-based participatory research (CBPR) approach, CIVIC will leverage: its long term relationships with the communities involved, an established CBPR Steering Committee developed and the knowledge gained as a Community Engagement Alliance (CEAL) grant recipient, the resources and networks of the University of Michigan CTSA (MICHR), and the expertise of our academic partners to identify and understand factors that contribute to COVID-19 vaccine hesitancy in African Americans and Latinx communities in Michigan. The investigators will develop and test interventions based on community-centered approaches to achieve a primary goal of increased vaccine uptake.

The investigators will achieve this goal with the following aims:

1. Increase understanding of the barriers and drivers of vaccine uptake and hesitancy;
2. Increase vaccine uptake and decrease vaccine hesitancy through the implementation and evaluation of a multi-component intervention; and maintain, enhance, and evaluate the effectiveness of the CIVIC partnership to equitably engage all partners.

DETAILED DESCRIPTION:
Like many states across the country, COVID-19 cases and deaths have impacted communities of color in Michigan at disproportionately higher rates than whites. A staggering reality is that while African Americans represent only 13.6% of Michigan's population, they represent 40% of the deaths from COVID-19.

* Half of the cases and deaths in Michigan occurred in Wayne County.
* Other Counties in the lower half of Michigan have similar disparities including Genesee, Washtenaw, and Kent.
* In Genesee County, where African Americans represent 20.3% of the population, they represent 35% of COVID-19 cases and 45% of deaths.
* In Washtenaw County, nearly half of the cases to date are located in two majority low-income zip codes in the city of Ypsilanti. African American residents, who make up 12% of the Washtenaw population, disproportionately constitute more than a quarter of the cases.
* And in Kent County, while 10.8% of the population is Latinx, this ethnic group makes up 32.4% of COVID-19 cases.

Preliminary data from the state reveal that these disparities will likely worsen due to significant hesitancy, fear, mistrust and misinformation regarding the COVID-19 vaccine if nothing is done to change current trends.

ELIGIBILITY:
Eligibility inclusion criteria:

* unvaccinated or unboosted adults 18 years and older who are interested in participating in the study OR vaccinated and boosted adults 18 years and older who are interested in becoming a Champion.
* Must be able to read and write in English or Spanish
* Must be able to receive SMS/MMS/text messages

Exclusion criteria:

* Persons under the age of 18
* unable to read or write English or Spanish
* unable or unwilling to receive SMS/MMS
* unwilling to consent
* for vaccine champions-unwillingness to complete communication trainings in English

No specific racial, ethnic, nor sex/gender group is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2025-09-11 (Estimated); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Self-reported COVID-19 Vaccine uptake | 6 months after the start of the intervention
  The primary outcome is the binary variable of participant-reported vaccine uptake over the 6 month intervention period. Participants will also be asked which vaccine, how many doses completed, location it was delivered, and date of delivery.

SECONDARY OUTCOMES:
Intention to uptake COVID-19 Vaccine | change from baseline at 6 months
  Vaccine Intentions will be assessed by asking, on a scale of 0-10, "how likely is it that you will get the COVID-19 vaccine?", with 0 being very unlikely and 10 being very likely. This will be analyzed using linear regression as described in the data analysis section.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Resnicow, Ph.D., Principal Investigator — University of Michigan; Emerson Delacroix, M.A.C.P., Study Director — University of Michigan; Erica Marsh, M.D., Principal Investigator — University of Michigan - Michigan Medicine
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
A deidentified dataset will be made available at the conclusion of the study per funder requirements.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The study team at the University of Michigan will disseminate the protocol with any deviations or adverse events to the UM-IRB. Data will be de-identified after the intervention phase ends which is planned for May 2024.
Access Criteria: The study team members will have access to the data and results at the end of the study.

DOCUMENTS (2):
  • Study Protocol (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT05096260/Prot_002.pdf
  • Informed Consent Form (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT05096260/ICF_001.pdf